CLINICAL TRIAL: NCT00504244
Title: A Randomized, Multicenter Study to Assess the Efficacy on Diseases Activity of Enteric-coated Mycophenolate Sodium Versus Continuation of Azathioprine in Patients With Systemic Lupus Erythematosus on Azathioprine Maintenance Therapy.
Brief Title: Myfortic Versus Azathioprine in Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Erasmus Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: P.L.A. van Daele, Erasmus MC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080ANL07
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; SLEDAI; Azathioprine; Myfortic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Mycophenolic Acid; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: switch to Myfortic — Myfortic 2 dd 720 mg
  Other Names: Myfortic
Drug: continuation of azathioprine — Azathioprine 2 mg/kg
  Other Names: Azathioprine

SUMMARY:
This study is designed to explore the use of myfortic ® in patients with active lupus erythematosus. Similar drugs in this class are increasingly used in organ transplantation and in autoimmune diseases. With the established safety profile of myfortic ® in allo-transplantation and the already existing data of mycophenolate mofetil in autoimmune diseases, this study should help to demonstrate the beneficial effect of myfortic ® on lupus activity. The aim of the study will be to show a decreased disease activity with myfortic ® compared to standard maintenance therapy with azathioprine.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a complex and potentially life-threatening disease that affects about 40 per 10,000 people in the general population (Mills 1994, Brown & Schrieber 1996). SLE is a chronic inflammatory disease characterized by auto-antibody overproduction and other distinct immunological abnormalities (Boumpas, et al 1995, Mohan & Datta 1995). It may affect the skin, joints, lungs, heart, serous membranes, nervous system or other organs. Improvements in treatment over the last decade have increased 10-year survival rates in Western countries to 90% or more, and 20-year survival rates of nearly 70% have also been reported (Abu-Shakra, et al 1995).

Newer treatment strategies include the use of novel immunosuppressive agents, such as mycophenolate mofetil (MMF). MMF has been widely used in solid-organ transplantation (Sollinger 1995, The Tricontinental Mycophenolate Mofetil Renal Transplantation Study Group 1996). MMF also has been used increasingly in autoimmune diseases (e.g., dermatomyositis, primary glomerular disease or psoriasis (Epinette, et al 1987, Gelber, et al 2000, Choi, et al 2002)).

MMF is the morpholinoethylester prodrug of mycophenolic acid (MPA). After oral administration MMF is well absorbed and rapidly hydrolyzed to MPA. MPA is a noncompetitive inhibitor of inosine monophosphate (IMP) dehydrogenase (DH). Inhibition of IMPDH leads to the depletion of deoxyguanosine triphosphate and a consequent decrease in the level of substrate required for DNA polymerase activity. This results in inhibition of DNA production and cell proliferation. T and B cells are more dependent on this de novo pathway of purine synthesis because alternative salvage pathways are unavailable. Thus, MPA is a selective inhibitor of lymphocyte proliferation, especially in activated lymphocytes (Allison & Eugui 2000).

A limited number of clinical studies have been performed to study the efficacy of MMF in the treatment of SLE. Most of these studies involved the treatment of nephritis. Chan, et al (2000) showed that the combination of MMF and prednisolone is as effective as a regimen of cyclophosphamide and prednisolone followed by azathioprine and prednisolone. Azathioprine and MMF as maintenance therapy were compared to cyclophosphamide therapy (Contreras, et al 2004) and appeared to be more efficacious and safer than long-term therapy with i.v. cyclophosphamide. In this study, it was also noted that patients treated with MMF had received lower doses of corticosteroids during maintenance therapy as compared to patients treated with azathioprine.

Recent reports suggest that MMF may also be effective in systemic lupus without severe renal involvement.(Pisoni, et al 2005) Yet, the superiority over azathioprine in this patient group has not been established. Own observations show that approximately 50% of patients with SLE treated with azathioprine have at least some evidence of lupus activity. The aim of this study will be to show a decreased lupus activity in patients treated with myfortic ® compared to therapy with azathioprine. Data so gathered may be useful in planning future developments in this indication

This is a 12 months, multi-center, 2-treatment arm, parallel-group, randomized, open label study in patients with systemic lupus erythematosus currently on azathioprine. The patients will be randomized to one of the following two treatment groups:

* Maintenance of previous therapy including azathioprine.
* Switch to a myfortic ® based regimen: myfortic ® (dose of 1440mg/day) A total of 48 patients (24 patients per arm) fulfilling the inclusion/exclusion criteria will be enrolled in the study from approximately 5 centers in the Netherlands. Screening evaluations and assessments will be performed in the period after informed consent has been signed by the patient and before randomization of the patient (Baseline, Day 1). Visits are scheduled for Baseline, Weeks 2, 4, 12, Months 6, 9 and 12.

The final analysis will be performed after the last patient has reached the 12 months of the study.

The following efficacy variables will be obtained and recorded:

* Disease activity index measured with SLEDAI
* Disease activity index measured with BILAG (numerical score)
* (Average) daily dose of prednisone (mg/kg/day). The dose will be measured from the patient starting the study and for the whole duration of the study.
* Damage index measured with SLICC/ACR
* Serum creatinine
* Creatinine clearance
* Urine protein:creatinine ratio

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged 18 years and over
* Patients meeting the diagnostic criteria for SLE (Appendix 2), according to ACR guidelines (including screening for anti-dsDNA (antibody to native DNA in abnormal titer))
* SLEDAI > 6
* Patients treated with maintenance therapy including azathioprine.
* Patients who are willing and able to participate in the study and from whom written informed consent has been obtained

Exclusion Criteria:

* Creatinine clearance of < 20ml/min
* Patients with any clinically significant infection
* Patients with known hypersensitivity to myfortic ® or to drugs with similar chemical structures
* Patients with a history of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin
* Patients with SLE active CNS manifestations or a past history of SLE CNS complications (e.g. psychosis, grand mal seizures)
* Patients who have received prior therapy with mycophenolic acids (MPAs) (e.g. MMF)
* Patients who have received an investigational drug within four weeks prior to study entry
* Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
SLEDAI | 12 months

SECONDARY OUTCOMES:
BILAG | 12 months
renal function | 12 months
Prednisone dose | 12 months
Quality of life (SF36) | 12 months
infections and side effects | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul LA van Daele, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- [Background] Allison AC, Eugui EM. Mechanisms of action of mycophenolate mofetil in preventing acute and chronic allograft rejection. Transplantation. 2005 Oct 15;80(2 Suppl):S181-90. doi: 10.1097/01.tp.0000186390.10150.66. PMID 16251851
- [Background] Chan TM, Tse KC, Tang CS, Mok MY, Li FK; Hong Kong Nephrology Study Group. Long-term study of mycophenolate mofetil as continuous induction and maintenance treatment for diffuse proliferative lupus nephritis. J Am Soc Nephrol. 2005 Apr;16(4):1076-84. doi: 10.1681/ASN.2004080686. Epub 2005 Feb 23. PMID 15728784
- [Background] Pisoni CN, Karim Y, Cuadrado MJ. Mycophenolate mofetil and systemic lupus erythematosus: an overview. Lupus. 2005;14 Suppl 1:s9-11. doi: 10.1191/0961203305lu2111oa. PMID 15803925
- [Background] Bombardier C, Gladman DD, Urowitz MB, Caron D, Chang CH. Derivation of the SLEDAI. A disease activity index for lupus patients. The Committee on Prognosis Studies in SLE. Arthritis Rheum. 1992 Jun;35(6):630-40. doi: 10.1002/art.1780350606. PMID 1599520
- [Background] Abu-Shakra M, Lee P. Mortality in systemic sclerosis: a comparison with the general population. J Rheumatol. 1995 Nov;22(11):2100-2. PMID 8596151
- [Background] Boumpas DT, Austin HA 3rd, Fessler BJ, Balow JE, Klippel JH, Lockshin MD. Systemic lupus erythematosus: emerging concepts. Part 1: Renal, neuropsychiatric, cardiovascular, pulmonary, and hematologic disease. Ann Intern Med. 1995 Jun 15;122(12):940-50. doi: 10.7326/0003-4819-122-12-199506150-00009. PMID 7755231
- [Background] Contreras G, Pardo V, Leclercq B, Lenz O, Tozman E, O'Nan P, Roth D. Sequential therapies for proliferative lupus nephritis. N Engl J Med. 2004 Mar 4;350(10):971-80. doi: 10.1056/NEJMoa031855. PMID 14999109
- [Background] Hay EM, Bacon PA, Gordon C, Isenberg DA, Maddison P, Snaith ML, Symmons DP, Viner N, Zoma A. The BILAG index: a reliable and valid instrument for measuring clinical disease activity in systemic lupus erythematosus. Q J Med. 1993 Jul;86(7):447-58. PMID 8210301
- [Background] Mills JA. Systemic lupus erythematosus. N Engl J Med. 1994 Jun 30;330(26):1871-9. doi: 10.1056/NEJM199406303302608. No abstract available. PMID 8196732
- [Background] Stoll T, Stucki G, Malik J, Pyke S, Isenberg DA. Association of the Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index with measures of disease activity and health status in patients with systemic lupus erythematosus. J Rheumatol. 1997 Feb;24(2):309-13. PMID 9034988